CLINICAL TRIAL: NCT00899964
Title: Influence of a Combined Personal and IT-based Physical Activity Intervention in an Obese, Sedentary Population on Daily Activity and Metabolic Risk Profile
Brief Title: IT-based Training in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2372/09
Record Dates: First submitted 2009-05-05; First posted 2009-05-12 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Obesity; Inactivity
MeSH Terms: conditions — Obesity; Sedentary Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): automated tailored feedback per E-mail
  Interventions: Behavioral: Physical activity
- 2 (Active Comparator): 1 + active contact per E-mail possible
  Interventions: Behavioral: Physical activity
- 3 (Active Comparator): 2 + active contact by trainer in case of exercise-related problems
  Interventions: Behavioral: Physical activity
- 4 (Active Comparator): 3 + regular active contact by trainer
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — 6-month physical activity intervention (endurance activities) delivered by internet with tailored training schedules

SUMMARY:
Though possibly cost-saving, there is little scientific evidence for the effectiveness and reasonable modality of internet-delivered physical activity interventions in primary prevention. The aim of the study is to compare the influence of different personal and IT-based service levels on the activity outcome of obese, sedentary persons to evaluate the minimum level of service necessary for a maximum increase in activity and weight reduction.

ELIGIBILITY:
Inclusion Criteria:

* Physical activity of less than once per week
* Body-Mass-Index 28-35 kg/m2
* Age 35-65
* Men and women

Exclusion Criteria:

* CHD
* Diabetes
* Other chronic diseases with conditions prohibiting regular physical activity
* Drug abuse
* BMI < 28 or > 35
* Regular physical activity
* Pregnancy
* Mental illness

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Self-reported physical activity evaluated by questionnaire | 6 months

SECONDARY OUTCOMES:
Body-Mass-Index | 6 months
Body weight | 6 months
Technology acceptance evaluated by questionnaire | 6 months
Motivation analysis | 6 months
Time spent on the internet | 6 months
Metabolic equivalents | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Prevention and Sports Medicine, München, Bavaria, Germany

REFERENCES:
- [Background] Bretschneider, U.; Ebner, W.; Leimeister, J. M.; Krcmar, H. (2007): Internetbasierte Ideenwettbewerbe als Instrument der Integration von Kunden in das Innovationsmanagement von Software-Unternehmen. In: Virtuelle Organisationen und Neue Medien 2007 /Workshop GeNeMe 2007: Gemeinschaften in neuen Medien. Herausgeber / Editor: Engelien, M.; Homann, J. Erscheinungsort / Published in: Lohmar, Köln Erscheinungsjahr / Year: 2007 Verlag / Publisher: Joseph Eul Verlag
- [Background] Dannecker, A., Konana, P., Leimeister, J. M.; Rajagopalan, B. (2007): Towards a Research Agenda for Virtual Communities. In: Proceedings of the Americas Conference on Information Systems (AMCIS 2007), Keystone
- [Background] Esch, S.; Knebel, U.; Leimeister, J. M.; Krcmar, H.: Referenzmodell für einen IT-gestützten mobilen Gesundheitscoach. In: Mobiles Computing in der Medizin, Proceedings zum 7. Workshop der GMDS-Arbeitsgruppe Mobiles Computing in der Medizin. Herausgeber: Leimeister, J.M.; Mauro, C.; Krcmar, H.; Eymann, T.; Koop, A., Shaker Verlag, Aachen, 2007
- [Background] Hörmann, C.; Klapdor, S.; Leimeister, J. M.; Krcmar, H. (2007): IT-Management in deutschen Kranken-häusern - eine empirische Untersuchung unter IT-Entscheidern. Arbeitspapier Nr. 27, Lehrstuhl für Wirtschaftsinformatik, Technische Universität München, März 2007
- [Background] Hoffmann, H.; Leimeister, J. M.; Krcmar, H. (2007): A Framework for Developing Personalizeable Mobile Services in Automobiles. In: XVth European Conference on Information Systems (ECIS 2007). Hrsg.: Österle, H.; Schelp, J.; Winter, R. University of St. Gallen, St. Gallen 2007, S. 938-949
- [Background] Hoffmann, H.; Leimeister, J. M.; Krcmar, H. (2007): Automotive Service Engineering - Systematische Entwicklung personalisierbarer und interaktiver mobiler Dienste für den Automobilsektor In: Proceedings of Wirtschaftsinformatik 2007 (Vol. 1), Universitätsverlag Karlsruhe, Karlsruhe 2007, S. 327-344
- [Background] Hoffmann, H., Leimeister, J. M., Krcmar, H. (2007): Pilotierung mobiler Dienste im Automobilsektor. In: Mobile Dienste im Auto der Zukunft. Hrsg. / Editors: Reichwald, R., Krcmar, H., Reindl, S. Publisher / Verlag: Eul-Verlag, Erscheinungsort / Published in: Lohmar, Erscheinungsjahr / Year: 2007, Seiten / Pages: 125-203
- [Background] Knebel, U.; Leimeister, J. M.; Krcmar, H. (2007): Personal Mobile Sports Companion: Design and Evaluation of IT-supported Product-Service-Bundles in the Sports Industry. In: XVth European Conference on Information Systems (ECIS 2007). Hrsg.: Österle, H.; Schelp, J.; Winter, R. University of St. Gallen, St. Gallen 2007, S. 81-92
- [Background] Leimeister, J. M.; Knebel, U.; Krcmar, H. (2007): Exploring Mobile Information Systems for Chronically Ill Adolescent Patients. In: International Journal of Web-based Communities (IJWBC), Ausgabe / Number: 4, Vol. 3, Verlag / Publisher: Inderscience, Erscheinungsjahr / Year: 2007
- [Background] Mauro, Ch.; Schweiger, A.; Sunyaev, A.; Leimeister, J. M., A., Krcmar, H. (2007): Single Sign-On Clinic Card-Lösung - Ein Konzept zur zentralen Verwaltung von Gesundheitskarten im stationären Umfeld. In: Proceedings of Informatik 2007, Bremen, GI - Gesellschaft für Informatik, S. 463-468
- [Background] Schweiger, A.; Leimeister, J. M.; Krcmar, H. (2007): Auf dem Weg zur integrierten Versorgungim Gesundheitswesen am Beispiel Krankenhaus: Parallelen aus Sicht der Wirtschaftsinformatik. In: Wissens-management im Krankenhaus. Hrsg. / Editor: Bohnet-Joschko, S. Publisher / Verlag: DUV - Gabler Edition Wissenschaft., Erscheinungsort / Published in: Wiesbaden, Erscheinungsjahr / Year: 2007, Seiten / Pages: 97-110
- [Background] Schweiger, A.; Sunyaev, A.; Leimeister, J. M.; Krcmar, H. (2007): Toward Seamless Healthcare with Software Agents. In: Communications of the Association for Information Systems (CAIS), Vol. 19, Verlag / Publisher: Association for Information Systems, Erscheinungsjahr / Year: 2007. Seiten / Pages 692-709
- [Background] Sunyaev, A.; Leimeister, J. M.; Schweiger, A.; Krcmar, H. (2007): Die elektronische Gesundheitskarte und die Sicherheit: Ein Vorschlag zur entwicklungsbegleitenden Sicherheitsevaluation aus Anwendersicht. In: Proceedings of Informatik 2007, Bremen, GI - Gesellschaft für Informatik, S. 469-474
- [Background] Veith, V.; Leimeister, J. M.; Krcmar, H. (2007): Towards Value-based Management of Flexible IT Envi-ronments. In: XVth European Conference on Information Systems (ECIS 2007). Hrsg.: Österle, H.; Schelp, J.; Winter, R. University of St. Gallen, St. Gallen 2007, S. 1190-1201
- [Background] Köbler, F.; Leimeister, J.M.; Lugmayr, A. (2006): Framework for Systematic and Strategic Planning of Innovation-based Mobile Broadband Services. Paper presented at the 14th Euromicro International Conference on Parallel, Distributed, and Network-Based Processing (PDP'06), Montbéliard, France
- [Background] Leimeister, J.M., Krcmar, H. (2006): Community Engineering - Systematischer Aufbau und Betrieb Virtueller Communities im Gesundheitswesen In: Wirtschaftsinformatik, Ausgabe / Number: 6, Vol. 48, Verlag / Publisher: Vieweg, Erscheinungsjahr / Year: 2006, Seiten / Pages 418-429
- [Background] Leimeister, J.M.; Krcmar, H. (2006): Designing and Implementing Virtual Patient Support Communities: A German Case Study In: The Internet and health care: Theory, research and practice. Hrsg. / Editors: Murero, M.; Rice, R.E. Publisher / Verlag: Lawrence Erlbaum Associates, Erscheinungsort/ Published in: Mahwah. Erscheinungsjahr / Year: 2006
- [Background] Leimeister, J. M.; Krcmar, H. (2006): Technologien für Online-Communities. In: Unternehmenskommunikation. Hrsg. / Editors: Muth, M.; Weidner, L.; Zehetbauer, E. Publisher / Verlag: Symposion Publishing, Erscheinungsort / Published in: Duesseldorf. Erscheinungsjahr / Year: 2006, Seiten / Pages: 1-14
- [Background] Neil, L.; Hansen, D.; Lindgaard, G.; Kogan, S.; Leimeister, J.M.; Oakley, K.; Selker, T. (2006): SIG Online Health Communities. Proccedings of the Conference on Human Factors in Computer Systems (CHI 2006), Montreal, S. 445
- [Background] Sandner, U.; Leimeister, J.M.; Krcmar, H. (2006): Business Potentials of Ubiquitous Computing. In: Managing Development and Application of Digital Technologies. Hrsg. / Editors: Kern, E.; Hegering, H.; Brügge, B. Publisher / Verlag: Springer, Erscheinungsort / Published in: Berlin. Erscheinungsjahr / Year: 2006, Seiten / Pages: 277-292
- [Background] Schweiger, A.; Leimeister, J.M.; Niggemann, J.; Feussner, H.; Krcmar, H. (2006): Softwareagenten für die Überwindung von Medienbrüchen bei der Patientenversorgung. In: HMD - Praxis der Wirtschaftsinformatik, Ausgabe / Number: 251, Vol. 43, Verlag / Publisher: dPunkt Verlag, Erscheinungsjahr / Year: 2006, Seiten / Pages 88-100